CLINICAL TRIAL: NCT03851900
Title: A Comparison of Long-Term Effectiveness of Two Desensitizing Products: A Randomized Clinical Placebo-Controlled Study
Brief Title: A Comparison of Long-Term Effectiveness of Two Desensitizing Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kerimova, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hacettepe 2017/06-26 KA-16009
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin hypersensitivity; Randomized clinical trial; Calcium phosphate desensitizer; Adhesive resin; VAS
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: For each patient, selected teeth will be randomly assigned to TM, SE or placebo by the lottery method. The subjects will blind to the agent being used. All applications will be performed by the same examiner.
Who Masked: Participant, Investigator
Masking Description: The subjects will blind to the agent being used. At each recall the investigator used blank sheets with patients' names only to avoid bias relative to previous assessments
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teethmate Desensitizer (TM) (Experimental): Calcium phosphate biomimetic material that forms hydroxyapatite from tetracalcium phosphate and dicalcium phosphate anhydrous and plug the dentin tubules causing remineralization and dentin hypersensitivity relief.
  Interventions: Other: Teethmate Desensitizer (TM)
- Clearfil SE Bond 2 (SE) (Active Comparator): Two-step self etch adhesive resin treating dentin hypersensitivity b covering a film layer after light-curing.
  Interventions: Other: Clearfil SE Bond 2
- Distilled water (Placebo Comparator): Distilled water with no desensitizing components.
  Interventions: Other: Distilled water

INTERVENTIONS:
Other: Teethmate Desensitizer (TM) — Desensitizing agent will be applied to sensitive teeth.
  Arms: Teethmate Desensitizer (TM)
Other: Clearfil SE Bond 2 — Desensitizing agent will be applied to sensitive teeth.
  Arms: Clearfil SE Bond 2 (SE)
Other: Distilled water — Placebo will be applied to sensitive teeth as a negative control.
  Arms: Distilled water

SUMMARY:
This randomized, controlled, clinical trial aimed to compare the 6- month clinical performance of a desensitizer that contains calcium phosphate TM with a two-step self-etch adhesive SE and placebo (distilled water). At least 150 teeth wil be treated with desensitizing products and placebo randomly one third usig TM, one third using SE and one third using placebo. The efficiency of the materials will be evaluated at baseline, 1 week, 1 month, 3 months and 6 months after treatment.

DETAILED DESCRIPTION:
The aim of this randomized, controlled, clinical trial is to compare the clinical efficacy of a desensitizer that contains calcium phosphate with a two-step self-etch adhesive and placebo through a long-term period (6 months). At least fifty patients with a sensitivity score of 6 or higher, according to the Visual Analog Scale (VAS), with at least three teeth will participate in this study. Teethmate Desensitizer (TM), Clearfil SE Bond 2 (SE) and placebo (distilled water) will be applied randomly to three teeth of each patient. Recalls will be done at baseline, 1 week, 1 month, 3 months and 6 months after treatment by applying air-blast and the sensitivity scores will be determined according to VAS. The efficiency of the materials will be determined according to the VAS scores. Data will be analyzed using Paired t test and repeated measures of ANOVA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with 3 or more hypersensitive teeth with a VAS (Visual Analog Scale) score
2. Willingness to participate in the study

Exclusion Criteria:

1. Subjects are unwilling to participate voluntarily
2. Patients under 18 years old
3. Those that were taking analgesic medicaments
4. Pregnant and breastfeeding females
5. The presence of a systemic disease that affects the participation
6. Teeth with cervical loss of hard tissue that need restoration absolutely
7. Large/defective restoration, caries or enamel cracks in sensitive teeth
8. Teeth with vulnerability to hypersensitivity after root scaling
9. Pulpitis presence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
The effectiveness of desensitizers through long-term period | 6 months
  The clinical efficacy of a desensitizer that contains calcium phosphate with a two-step self-etch adhesive and placebo through a long-term period. Evaluation will be performed usig the Visual Analog Scale(VAS). VAS values will be according to the following parameters: 0 - no discomfort;1 to 3 - light discomfort;4 to 6 - mild discomfort;7 to 9 - severe discomfort;10 - Unbearable discomfort. After each stimulus to the suspected site the degree of hypersensitivity will be determined from 6 to 10 as the preop VAS score for each individual painful tooth.

SECONDARY OUTCOMES:
Subjective satisfaction of patients | 6 months
  Because of the patient-centered aspect of the study patients' subjective satisfaction will be prior. Patients will be asked to define their sensitivity according to Visual Analog Scale (VAS) scale. VAS values will be according to the following parameters:
  0 - no discomfort;1 to 3 - light discomfort;4 to 6 - mild discomfort;7 to 9 - severe discomfort;10 - Unbearable discomfort. In case of persistant or recurrent sensitivity reported by the participants after application of desensitizing agents or placebo, even if the Visual Analog Scale score was decreased, it was accepted as failure, so alternative hypersensitivity treatments applied and current teeth will be excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Arlin Kiremitci, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)